CLINICAL TRIAL: NCT04849052
Title: A Randomized Pilot Trial of a Multicomponent Interactive Text Message Intervention to Promote Physical Activity in Midlife Adults
Brief Title: Text Messaging to Increase Activity in Midlife
Acronym: MASTERY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021P000881
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Middle Aged
Keywords: Text Message; Physical Activity; Stress Reduction; Positive Psychology; Well-being
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blinded study
Who Masked: Outcomes Assessor
Masking Description: While participants and study trainers will be aware of group assignment, a blinded study team member will perform outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASTERY Intervention (Experimental): Participants will complete a positive psychology activity, work towards a physical activity goal, and use a stress reduction technique, then will complete weekly text message sessions. In the first six weeks, participants will review the activities they performed the prior week, be introduced to new material, choose activities to perform that week, and set a new physical activity goal during the text message sessions. In the final 6 weeks, participants will review progress towards prior goals, set new physical activity goals, and choose positive psychology and stress reduction skills to use that week. Finally, over the course of the program participants will complete three brief calls with a study trainer to discuss progress.
  Interventions: Behavioral: MASTERY
- Attentional control (Active Comparator): Participants will receive the same physical activity component noted in MASTERY along with added messages providing education and guidance about physical activity, from our past work. Control participants will not receive PP or midlife-related content.
  Interventions: Behavioral: Attentional Control

INTERVENTIONS:
Behavioral: MASTERY — In MASTERY, participants will have interactive, two-way text message 'sessions' (5-10 minutes of two-way text communication with an automated text-message program) once weekly for 12 weeks. Furthermore, study trainers will conduct 4 brief calls with participants (Weeks 1, 4, 7, and 12) to introduce the program, assess progress, answer questions, and provide support.
  Arms: MASTERY Intervention
Behavioral: Attentional Control — Participants in the control condition will also receive text messages once per week. To ensure time matching, the program will have 4 phone check-ins (on physical activity) as in MASTERY.
  Arms: Attentional control

SUMMARY:
This is a randomized controlled pilot trial of a text message intervention to promote physical activity in midlife adults (MASTERY), compared to an attention-matched control condition. The MASTERY intervention utilizes two-way text message sessions once-weekly for 12 weeks focusing on performing activities to enhance well being, setting physical activity goals, and learning techniques to reduce midlife-specific stress.

DETAILED DESCRIPTION:
This is a randomized controlled pilot trial of a multipronged intervention to promote physical activity in midlife adults (MASTERY), compared to an attention-matched control condition. In MASTERY, participants will have interactive, two-way text message 'sessions' (5-10 minutes of two-way text communication with an automated text-message program) once weekly for 12 weeks. The messages will focus on 3 distinct areas in the same order each week: (1) well-being-based skills and assigned activities, customized for midlife adults, (2) physical activity content focused on setting and reaching weekly activity goals, and (3) specific skills to manage midlife-related stressors that act as barriers to activity. The primary outcome is objectively measured moderate to vigorous physical activity (MVPA). Secondary outcomes include feasibility and acceptability and other activity-related, psychological, and functional outcomes at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Midlife status (age 45-64 at enrollment).
2. Low baseline physical activity (≤150 minutes/week of MVPA]) as initially self-reported via the well-validated IPAQ and then confirmed via accelerometer after 7 days of wear.

Exclusion Criteria:

1. Existing coronary artery disease (CAD; diagnosed via cardiac catheterization using standard coronary artery stenosis definitions or prior ACS).
2. An unrelated condition limiting physical activity (e.g., ambulation with a cane or walker, recent or planned surgery, or other condition such that ability to increase moderate to physical activity would be limited).
3. Participation in any other programs focused on cardiac prevention or well-being (e.g., cardiac rehabilitation).
4. A cognitive disturbance precluding participation or informed consent, assessed using a six-item screen7 designed to assess suitability for research participation.
5. Inability to speak/write fluently in English.
6. No access to a text message-capable phone.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Moderate-Vigorous Physical Activity [MVPA] | Baseline, 6 weeks, 12 weeks
  ActiGraph accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline, 6 weeks, and 12 weeks. We will report change from baseline to 6 weeks and 12 weeks in the average number of minutes of MVPA performed per day.

SECONDARY OUTCOMES:
Proportion of text message sessions completed | Weekly over 12 weeks.
  To assess the feasibility of the MASTERY intervention the automated platform will record rates of the proportion of text message sessions in which participants respond and set a physical activity goal.
Mean utility ratings of positive psychology text messages | 6 weeks; 12 weeks
  Participants will rate the utility of the positive psychology text message sessions over the past six weeks on a scale of 0 (unhelpful) to 10 (very helpful).
Mean utility ratings of physical activity text messages | 6 weeks; 12 weeks
  Participants will rate the utility of the physical activity text message sessions over the past six weeks on a scale of 0 (unhelpful) to 10 (very helpful).
Mean utility ratings of stress reduction text messages | 6 weeks; 12 weeks
  Participants will rate the utility of the stress reduction text message sessions over the past six weeks on a scale of 0 (unhelpful) to 10 (very helpful).
Mean utility ratings of phone check-ins | 6 weeks; 12 weeks
  Participants will rate the utility of the phone sessions over the past six weeks on a scale of 0 (unhelpful) to 10 (very helpful).
Change in overall physical activity | Baseline, 6 weeks, 12 weeks
  ActiGraph accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline, 6 weeks, and 12 weeks. We will report change from baseline to 6 weeks and 12 weeks in the average number of steps per day.
Change in sedentary leisure time | Baseline, 6 weeks, 12 weeks
  ActiGraph accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline, 6 weeks, and 12 weeks. We will report change from baseline to 6 weeks and 12 weeks in the average number of minutes of sedentary leisure time per day. Participants will indicate which hours represent leisure time during workdays and off days/weekends to allow us to ascertain this outcome.
Change in self-reported physical activity | Baseline, 6 weeks, 12 weeks
  The International Physical Activity Questionnaire (IPAQ) is a well-validated 7-day physical activity recall assessment for physical activity. Activity will be measured by the number of MET-minutes of moderate or greater activity per week, and change will be assessed by subtracting the baseline score from the 6- and 12-week scores.
Change in positive affect (positive affect items of the Positive and Negative Affect Schedule [PANAS]) | Baseline, 6 weeks, 12 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of positive affect.
Change in optimism (Life Orientation Test - Revised [LOT-R]) | Baseline, 6 weeks, 12 weeks
  The Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of optimism.
Change in life satisfaction (Satisfaction with Life Scale [SWLS]) | Baseline, 6 weeks, 12 weeks
  The Satisfaction with Life Scale is a 5-item scale designed to measure global cognitive judgments of one's life satisfaction (Range: 5-35). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks.
Change in depressive symptoms (Hospital Anxiety and Depression Scale depression subscale [HADS-D]) | Baseline, 6 weeks, 12 weeks
  The Hospital Anxiety and Depression Scale depression subscale (HADS-D) will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of depression.
Change in anxiety (Hospital Anxiety and Depression Scale anxiety subscale [HADS-A]) | Baseline, 6 weeks, 12 weeks
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of anxiety.
Change in exercise self-efficacy (Self-efficacy for Exercise Scale [SES]) | Baseline, 6 weeks, 12 weeks
  The Self-efficacy for Exercise Scale will be used to measure exercise self-efficacy. This is a 9-item scale used to assess an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 20+ minutes per session in the future. (Range: 0-90). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of self-efficacy.
Change in social support (Norbeck Social Support Questionnaire) | Baseline, 6 weeks, 12 weeks
  The Norbeck Social Support Questionnaire will be used to assess an individual's perceived emotional and tangible support. Likert scale ratings for each person in the individual's social network will be made and the average across the social network will be calculated (Range:0-4). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of perceived social support.
Change in perceived constraints (perceived constraints subscale of the MIDUS Sense of Control measure) | Baseline, 6 weeks, 12 weeks
  The 8-item subscale of the MIDUS Sense of Control measure will be used to measure internal locus of control - perceived constraints (Range: 8-56). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of perceived constraints.
Change in personal mastery (personal mastery subscale of the MIDUS Sense of Control measure) | Baseline, 6 weeks, 12 weeks
  The 4-item subscale of the MIDUS Sense of Control measure will be used to measure internal locus of control - perceived constraints (Range: 4-28). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate higher levels of perceived constraints.
Change in function (General Health Questionnaire-12 [GHQ-12]) | Baseline, 6 weeks, 12 weeks
  The General Health Questionnaire-12 consists of 12 items and assesses function (Range: 0-36). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate worse functional status.
Change in mental health related quality of life (Medical Outcomes Study Short Form-12 mental component score [SF-12 MCS]) | Baseline, 6 weeks, 12 weeks
  Mental health related quality of life will be assessed via the mental component score of the Medical Outcomes Study SF-12 (Range: 0-100). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate better health-related quality of life.
Change in physical health related quality of life (Medical Outcomes Study Short Form-12 physical component score [SF-12 PCS]) | Baseline, 6 weeks, 12 weeks
  Physical health related quality of life will be assessed via the physical component score of the Medical Outcomes Study SF-12 (Range: 0-100). Change will be calculated by subtracting the score at baseline from the score at 6 and 12 weeks. Higher scores indicate better health-related quality of life.
Change in body weight | Baseline, 6 weeks, 12 weeks
  Body weight (in kilograms) will be measured by nurses. Change will be calculated by subtracting the weight at baseline from the weight at 6 and 12 weeks.
Change in body mass index (in kilograms per square meter) | Baseline, 6 weeks, 12 weeks
  Height and weight will be measured by nurses at baseline, 6, and 12 weeks. Change will be calculated by subtracting the baseline value from the value at 6 and 12 weeks.
Change in waist circumference (in centimeters) | Baseline, 6 weeks, 12 weeks
  Waist circumference will be measured by nurses at baseline, 6, and 12 weeks. Change will be calculated by subtracting the baseline value from the value at 6 and 12 weeks.
Change in blood pressure (millimeters of mercury) | Baseline, 6 weeks, 12 weeks
  Blood pressure will be measured by nurses at baseline, 6, and 12 weeks. Change will be calculated by subtracting the baseline value from the value at 6 and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No